CLINICAL TRIAL: NCT04282070
Title: A Phase Ib, Open-label Trial to Investigate the Safety and Tolerability of SHR-1701 in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Brief Title: SHR-1701 in Patients With Recurrent/Metastatic Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1701-I-103
Record Dates: First submitted 2020-02-18; First posted 2020-02-24 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-03

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — SHR-1701; Gemcitabine; Injections; Cisplatin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR-1701 (Arm A) (Experimental): SHR-1701 for R/M NPC failure after platinum-based chemotherapy
  Interventions: Drug: SHR-1701
- SHR-1701 (Arm B) (Experimental): SHR-1701 for R/M NPC failure after anti PD-1/PD-L1 antibody therapy
  Interventions: Drug: SHR-1701
- SHR-1701 plus Gemcitabine and Cisplatin (Arm C) (Experimental): SHR-1701+Gemcitabine+Cisplatin for first line treatment of R/M NPC
  Interventions: Drug: SHR-1701; Drug: Gemcitabine; Drug: Cisplatin
- SHR-1701 plus Albumin Paclitaxel (Arm D) (Experimental): SHR-1701+Albumin Paclitaxel for R/M NPC failure after first line anti PD-1/PD-L1 antibody therapy
  Interventions: Drug: SHR-1701; Drug: Albumin Paclitaxel

INTERVENTIONS:
Drug: SHR-1701 — Subjects will receive an intravenous infusion of SHR-1701 until confirmed progression, unaccepted toxicity, or any criterion for withdrawal from the trial.
  Other Names: SHR-1701 Injection
Drug: Gemcitabine — Maximum 6 cycles for combined therapy.
  Other Names: Gemcitabine Hydrochloride for Injection
  Arms: SHR-1701 plus Gemcitabine and Cisplatin (Arm C)
Drug: Cisplatin — Maximum 6 cycles for combined therapy.
  Other Names: Cisplatin Injection
  Arms: SHR-1701 plus Gemcitabine and Cisplatin (Arm C)
Drug: Albumin Paclitaxel — Maximum 6 cycles for combined therapy.
  Other Names: nab-Paclitaxel
  Arms: SHR-1701 plus Albumin Paclitaxel (Arm D)

SUMMARY:
This is an open label, phase Ib Study of SHR-1701 in patients with recurrent/metastatic nasopharyngeal carcinoma(R/M NPC).

DETAILED DESCRIPTION:
The main purpose of this study is to assess the safety and tolerability of SHR-1701 in patients with R/M NPC. The secondary purpose is to assess the anti-tumor activity and immunogenicity of SHR-1701 in R/M NPC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Recurrent/Metastatic Nasopharyngeal Carcinoma
* Subjects failure after platinum-based chemotherapy; failure from anti-PD-1/PD-L1 antibody therapy; Primarily metastatic (stage IVB as defined by the International Union against Cancer and American Joint Committee on Cancer staging system for NPC, eighth edition) or recurrent NPC that is not amenable for local regional treatment or curative treatment; failure from first line anti-PD-1/PD-L1 antibody therapy.
* Able and willing to provide signed informed consent form, and able to comply with all procedures.
* Histologically or cytologically proven metastatic or locally advanced solid tumors.
* Life expectancy >= 12 weeks as judged by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 at trial entry.
* Disease must be measurable with at least 1 uni dimensional measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Adequate hematological, hepatic and renal function as defined in the protocol Other protocol-defined inclusion criteria could apply.

Exclusion Criteria:

* Prior therapy with an anti-PD1, anti-PD-L1, anti-CTLA-4 or a TGFb inhibitor.
* Anticancer treatment within 28 days before the first dose of study drug.
* Major surgery within 28 days before start of trial treatment.
* Systemic therapy with immunosuppressive agents within 7 days prior to the first dose of study drug; or use any investigational drug within 28 days before the start of trial treatment.
* With any active autoimmune disease or history of autoimmune disease.
* With active central nervous system (CNS) metastases causing clinical symptoms or requiring therapeutic intervention.
* Clinically significant cardiovascular and cerebrovascular diseases
* History of immunodeficiency including seropositive for human immunodeficiency virus (HIV), or other acquired or congenital immunedeficient disease, or any active systemic viral infection requiring therapy.
* Previous malignant disease (other than the target malignancy to be investigated in the trial) within the last 2 years. Subjects with history of cervical carcinoma in situ, superficial or non-invasive bladder cancer or basal cell or squamous cell cancer in situ previously treated with curative intent are NOT excluded.
* Receipt of any organ transplantation, including allogeneic stem-cell transplantation Other protocol-defined exclusion criteria could apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-04-16 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
Toxicity Toxicity | up to 2 years
  Number of participants with adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per RECIST 1.1 | up to 2 years
  ORR is defined as the percentage of participants in the analysis population who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: at least 30% decrease in the sum of diameters of target lesions) per RECIST 1.1.
Progression-free Survival (PFS) per RECIST 1.1 | up to 2 years
  PFS is defined as the time from randomization to the first documented disease progression per RECIST 1.1 based on blinded independent central review or death due to any cause, whichever occurs first.
Disease Control Rate (DCR) per RECIST 1.1 | up to 2 years
  DCR is defined as the percentage of participants in the analysis population who have a CR, PR or SD per RECIST 1.1.
Immunogenicity of SHR-1701 | up to 2 years
  anti SHR-1603 antibodies (ADA)
Overall Survival (OS) | up to 2 years
  Overall Survival is defined as the time from registration to death due to any cause, or censored at date last known alive. OS will be measured by the Method of Kaplan and Meier.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of Guangzhou Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No